CLINICAL TRIAL: NCT00877292
Title: The RNA (RNA-Based Noninvasive Aneuploidy) Study
Brief Title: A New Prenatal Blood Test for Down Syndrome
Acronym: RNA
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Sequenom, Inc. (Industry)
Responsible Party: Principal Investigator, Glenn E. Palomaki PhD, Prinicpal Investigator, Women and Infants Hospital of Rhode Island
Other Study IDs: 09-0004
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Down Syndrome; Trisomy 21
Keywords: Down Syndrome; trisomy 21; prenatal testing; pregnant women
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fetal RNA and DNA in maternal plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Down syndrome: Women having CVS or amniocentesis who, as a group, have a high prevalence of Down syndrome.

SUMMARY:
The study will examine the sensitivity and specificity of a circulating cell-free nucleic acid test (DNA/RNA) to identify Down syndrome between about 10 weeks and 21 weeks 6 days gestation. In addition, the new test may be used to identify trisomy 13 and 18 as part of a more complete laboratory developed test. We hypothesize that the new circulating cell-free fetal NA-based test will accurately and precisely measure specific fetal markers in maternal circulation and that measurement will lead to the ability to noninvasively identify with high sensitivity and specificity, fetal chromosome abnormalities, such as Down syndrome.

DETAILED DESCRIPTION:
The RNA study is an observational trial whose primary aim is to document the performance (sensitivity and specificity) of one or more laboratory developed test (LDT) using circulating cell-free fetal nucleic acids from maternal plasma to identify Down syndrome. Multiple test modalities are being pursued, including massively parallel sequencing and those utilizing differential methylation. The population being studied is women already having a diagnostic test (e.g., amniocentesis, CVS) between 10 weeks and 21 weeks 6 days gestation, and whose pregnancy is at high risk for having Down syndrome. The women provide informed consent. The karyotype will provide the gold standard against which the LDT test is judged. Samples and karyotypes will be collected from up to 25 prenatal diagnostic centers around the world and tested in several laboratories in the United States. The secondary aim is to develop a nucleic acid sample bank to allow documentation of subsequent improvements or new methodologies to identify fetal aneuploidy using circulating cell-free fetal nucleic acids.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between about 10 weeks and 21 weeks 6 days gestation who are undergoing a diagnostic procedure (i.e., chorionic villus sampling or amniocentesis) for karyotype analysis who have, on average, a high prevalence of Down syndrome (about 1:30 to 1:50).
* Three main sources are pregnancies screen positive for:

  1. the combined test at 10 to 13 weeks (NT, PAPP-A and hCG)
  2. the second trimester quadruple test at 15 to 18 weeks gestation
  3. integrated screening (PAPP-A and the quadruple test, with or without NT).
* Variations of the integrated test such as sequential testing will also be acceptable.
* Other, less common high risk groups would be women having diagnostic testing because of maternal age of 38 years or older at delivery, pregnancies with an abnormal ultrasound highly suggestive of a chromosome abnormality (e.g., major heart defect, clenched fist), and women with an inherited form of Down syndrome (Robertsonian translocation).

Exclusion Criteria:

* Nonpregnant women and women at relatively low risk for a Down syndrome baby.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women between about 10 weeks and 21 weeks 6 days gestation who are undergoing a diagnostic procedure (i.e., chorionic villus sampling or amniocentesis) for karyotype analysis.
Sampling Method: Non-Probability Sample
Enrollment: 4664 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The RNA study is an observational trial whose primary aim is to document the performance (sensitivity and specificity) of a laboratory developed test (LDT), using fetal nucleic acid in maternal plasma to identify Down syndrome in early pregnancy. | Within 1st and 2nd trimesters

SECONDARY OUTCOMES:
The secondary aim is to develop a sample bank to allow documentation of subsequent improvements in the existing LDT or documenting performance of new methodologies. | Late1st and early 2nd trimesters

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O'Brien, MD, Principal Investigator — Women and Infants Hospital
Locations (27):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Northwestern University, FSM, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - New Beginnings Perinatal Consultants, Providence, Rhode Island
  - Women and Infants Hospital, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - Intermountain Health Care, Murray, Utah
  - UVA Medical Center, Charlottesville, Virginia
- Argentina (2):
  - Center for Medical Education and Clinical Investiagtion, Buenos Aires
  - Sociedad Italiana de Beneficencia en Buenos Aires - Hospital Italiano, Buenos Aires
- University of Sydney, St Leonards, New South Wales, Australia
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Children's and Women's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - North York General Hospital, Toronto, Ontario
- Czechia (2):
  - Imalab, Zlín, Zlín
  - Centrum lekarske genetiky s.r.o., České Budějovice
- Hungary (2):
  - Semmelweis University, Budapest
  - Pecs University, Pécs
- Rotunda Hospital, Dublin, Ireland
- Rambam Medical Center, Haifa, Israel
- U.O. Ostetricia e Ginecologia Laboratorio Sperimentale di Tecniche, Genova, Italy
- Hospital Clinic Barcelona - Maternitat Campus, Barcelona, Catalonia, Spain

REFERENCES:
- [Result] Palomaki GE, Deciu C, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma reliably identifies trisomy 18 and trisomy 13 as well as Down syndrome: an international collaborative study. Genet Med. 2012 Mar;14(3):296-305. doi: 10.1038/gim.2011.73. Epub 2012 Feb 2. PMID 22281937
- [Result] Canick JA, Kloza EM, Lambert-Messerlian GM, Haddow JE, Ehrich M, van den Boom D, Bombard AT, Deciu C, Palomaki GE. DNA sequencing of maternal plasma to identify Down syndrome and other trisomies in multiple gestations. Prenat Diagn. 2012 Aug;32(8):730-4. doi: 10.1002/pd.3892. Epub 2012 May 14. PMID 22585317
- [Result] Palomaki GE, Kloza EM, Lambert-Messerlian GM, van den Boom D, Ehrich M, Deciu C, Bombard AT, Haddow JE. Circulating cell free DNA testing: are some test failures informative? Prenat Diagn. 2015 Mar;35(3):289-93. doi: 10.1002/pd.4541. Epub 2015 Jan 8. PMID 25449554
- [Result] Lambert-Messerlian G, Kloza EM, Williams J 3rd, Loucky J, O'Brien B, Wilkins-Haug L, Mahoney MJ, De Biasio P, Borrell A, Ehrich M, van den Boom D, Bombard AT, Deciu C, Palomaki GE. Maternal plasma DNA testing for aneuploidy in pregnancies achieved by assisted reproductive technologies. Genet Med. 2014 May;16(5):419-22. doi: 10.1038/gim.2013.149. Epub 2013 Oct 3. PMID 24091801
- [Result] Mazloom AR, Dzakula Z, Oeth P, Wang H, Jensen T, Tynan J, McCullough R, Saldivar JS, Ehrich M, van den Boom D, Bombard AT, Maeder M, McLennan G, Meschino W, Palomaki GE, Canick JA, Deciu C. Noninvasive prenatal detection of sex chromosomal aneuploidies by sequencing circulating cell-free DNA from maternal plasma. Prenat Diagn. 2013 Jun;33(6):591-7. doi: 10.1002/pd.4127. PMID 23592550
- [Result] Canick JA, Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE. The impact of maternal plasma DNA fetal fraction on next generation sequencing tests for common fetal aneuploidies. Prenat Diagn. 2013 Jul;33(7):667-74. doi: 10.1002/pd.4126. Epub 2013 May 31. PMID 23592541
- [Result] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Derived] Palomaki GE, Ashwood ER, Best RG, Lambert-Messerlian G, Knight GJ. Is maternal plasma DNA testing impacting serum-based screening for aneuploidy in the United States? Genet Med. 2015 Nov;17(11):897-900. doi: 10.1038/gim.2015.39. Epub 2015 Apr 2. PMID 25834952
- [Derived] Kloza EM, Haddow PK, Halliday JV, O'Brien BM, Lambert-Messerlian GM, Palomaki GE. Evaluation of patient education materials: the example of circulating cell free DNA testing for aneuploidy. J Genet Couns. 2015 Apr;24(2):259-66. doi: 10.1007/s10897-014-9758-8. Epub 2014 Sep 10. PMID 25204423